CLINICAL TRIAL: NCT06310148
Title: An Evaluation of the Effectiveness and Cost-effectiveness of the Chronic Disease Co-Care (CDCC) Pilot Scheme: a Commissioned Study
Brief Title: Evaluation of the Chronic Disease Co-Care Pilot Scheme
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government); Primary Healthcare Office, Hong Kong (Unknown)
Responsible Party: Principal Investigator, Dr. Eric Yuk Fai Wan, Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UW 24-019
Record Dates: First submitted 2024-02-11; First posted 2024-03-15 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Chronic Disease; Disease Management; Primary Healthcare
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participating in Chronic Disease Co-Care Pilot Scheme (Experimental): Participants will receive comprehensive health management plans and necessary medication treatment from family doctors, based on their clinical condition. Nurse clinic will provide disease prevention education, health assessment, and counselling services, whereas allied health professionals (including optometrists, podiatrists, dietitians, and physiotherapists) will provide individualized intervention services for participants.
  Interventions: Combination Product: The Chronic Disease Co-Care (CDCC) Pilot Scheme
- Not participating in Chronic Disease Co-Care Pilot Scheme (No Intervention): Eligible non-CDCC participants will only be referred to the laboratories of a designated service provider by the research team for physical examination, blood tests, and urine test as a screening for DM and HT. No health management plans and necessary medication treatment would be provided to them in this study.

INTERVENTIONS:
Combination Product: The Chronic Disease Co-Care (CDCC) Pilot Scheme — Participants will receive comprehensive health management plans and necessary medication treatment from family doctors, based on their clinical condition. Nurse clinic will provide disease prevention education, health assessment, and counselling services, whereas allied health professionals (including optometrists, podiatrists, dietitians, and physiotherapists) will provide individualized intervention services for participants.
  Arms: Participating in Chronic Disease Co-Care Pilot Scheme

SUMMARY:
The Chronic Disease Co-Care (CDCC) Pilot Scheme is initiated for early screening and management of people with hypertension (HT), pre-diabetes mellitus (pre-DM) and diabetes mellitus (DM) in Hong Kong. This study will evaluate the quality of care, feasibility, acceptability, effectiveness and cost-effectiveness of the Scheme.

This is a 12-month cohort study among the District Health Centre (DHC) or DHC Express, healthcare providers, CDCC participants and a comparison group of 1,886 non-participants. All the person-in charge, 2 family doctors and 1 of each allied health provider from each DHC/DHC Express will be administered with the questionnaires on quality of care and costing. All CDCC participants will be included in subject characteristics, among which a convenience sample of 548 will complete a telephone survey on experience, enablement and satisfaction of the CDCC Pilot Scheme. The health outcomes of 1,886 CDCC participants and 1,886 non-participants will be compared for evaluation of effectiveness and cost-effectiveness.

Participant characteristics, enablement, compliance to the standards of care, and costing of CDCC Pilot Scheme will be summarized using descriptive statistics. Differences in the proportion of patients meeting treatment targeted for HT, pre-DM and DM after 12 months will be compared by chi-squared test and logistic regressions. The incremental cost-effectiveness ratio will be evaluated by comparing with the World Health Organization (WHO) threshold. This study will inform future healthcare planning and policy for manpower and resource allocation.

DETAILED DESCRIPTION:
This study aims to evaluate the quality of care, feasibility, acceptability, effectiveness and cost-effectiveness of the CDCC Pilot Scheme in Hong Kong. The objectives of this study are the following:

1. Describe the characteristics of participants of the CDCC Pilot Scheme;
2. Measure the standards of adherence to care criteria achieved by healthcare providers participating in the CDCC Pilot Scheme;
3. Evaluate participant acceptability by self-reported outcomes on enablement, experience and satisfaction level about the services of CDCC;
4. Evaluate the effectiveness of the CDCC Pilot Scheme on improving health outcomes among CDCC participants over 12 months;
5. Determine the provider costs and cost-effectiveness for delivering the CDCC Pilot Scheme relative to its effectiveness on participants health outcomes

The detailed study design of each objective are:

Objective (a): All participants in CDCC Pilot Scheme between 1 Jan 2024 and 30 Jun 2024 will be included in the evaluation. The characteristics including demographics, comorbidities, and medications of the participants will be summarized using descriptive statistics.

Objective (b): For the evaluation of the structure of care, quantitative data will be collected through structured questionnaires on the quality of care with DHC/DHC Express managers at 6 months and repeated at 12 months. Each DHC/DHC Express will also nominate two family doctors and one of each network allied health professionals (optometrists, podiatrists, dietitians, and physiotherapists subject to the availability in each center) within their service network to complete the questionnaire at 12 months. For the evaluation of the standards on process and outcome of care, all participants in the CDCC Pilot Scheme between 1 Jan 2024 and 30 Jun 2024 will be included.

Objective (c): Participants will be conveniently sampled after completion of the Health Risk Factor Assessment (HRFA) at DHC/DHC Express between 1 Jan 2024 and 31 Mar 2024 to complete surveys on self-reported outcomes. For the first survey at 3 months, a questionnaire will be used to assess participants' enablement level and experience during the screening phase. The second follow-up survey will be administered at 12 months to assess participants' experience in clinical encounters.

Objective (d): This will be a 1-year comparative cohort study including CDCC and non-CDCC participants to evaluate the effectiveness of the CDCC Pilot Scheme. A total of 264 CDCC participants, and 264 non-CDCC participants screened positive for HT, pre-DM, or DM will be included as intervention and comparison group, respectively. All participants will be followed up 12 months. Records for CDCC participants who meet the inclusion criteria between 1 Jan 2024 and 30 Apr 2024, will be extracted from the Electronic Health Record Sharing System database. Meanwhile, a convenient sample of 1,886 non-CDCC participants (comparison group) will be recruited from the community between 1 Jan 2024 and 30 Apr 2024.

Objective (e): This will be a 1-year comparative cohort study including CDCC and non-CDCC participants to evaluate the costs and cost-effectiveness of the CDCC Pilot Scheme. The total costs incurred on the CDCC Pilot Scheme from 1st January 2024 to 31st December 2024, including set-up costs, ongoing operational costs and ongoing administrative and maintenance costs will be collected via questionnaires. Direct medical costs for CDCC participants and non-CDCC participants will be collected after 12 months.

ELIGIBILITY:
Inclusion Criteria of interventional group:

* Hong Kong residents
* Aged ≥45 years
* Registered as a member of DHC/DHC Express
* Provided informed consent on sharing their data in the electronic Health Record Sharing System
* Provided consent to join the CDCC Pilot Scheme Terms and Conditions.

Exclusion Criteria of interventional group:

* With known history of DM or HT

Inclusion Criteria of comparison group:

* Hong Kong residents
* Aged ≥45 years
* Provided informed consent for the study.

Exclusion Criteria of comparison group:

* Without known history of DM or HT

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3772 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Characteristics of the Chronic Disease Co-Care (CDCC) participants | Characteristics of CDCC participants will be described at baseline
  Characteristics including demographics, comorbidities, and medications of the CDCC participants. For continuous variables, age will be presented in years, blood pressure will be presented in millimeters of mercury, fasting glucose, low-density-lipoprotein cholesterol and triglycerides will be presented in millimole per liter, weight in kilograms and height in meter will be combined to report body mass index (BMI) in kg/m^2, estimated glomerular filtration rate will be presented in milliliters per minute per 1.73m^2. For categorical variables, frequency and proportion will be used. participants. For continuous variables, age will be presented in years. For categorical variables, frequency and proportion will be used.
Healthcare providers' adherence to care standards on the evaluation framework by the quality of care questionnaire | Questionnaires will be implemented at 6 months and 12 months after the study begins
  The standards (proportion of participants) achieved by the program in each of the criterion specified under each domain of quality of care according to the CDCC Pilot Scheme protocol. The questionnaire is developed based on the evaluation framework on structure, process and outcome. The percentage of adherence out of 100% based on pre-determined key performance indicators will be reported. A higher score means a greater adherence to the standards of care.
Enablement of CDCC participants by the Chinese Patient Enablement Instrument | 12 months
  Participants' enablement will be measured by the Chinese Patient Enablement Instrument (PEI) at 12 months following the enrolment into the CDCC Pilot Scheme
Effectiveness of the CDCC Pilot Scheme on disease control for pre-diabetes mellitus (pre-DM) and DM in percent of Glycated Hemoglobin (HbA1c) and hypertension (HT) in millimeter of mercury of systolic blood pressure (SBP)/diastolic blood pressure (DBP) | 12 months
  Differences in the proportion of CDCC participants achieving the target outcome of disease control after 12 months as compared with non-CDCC participants. Target outcomes of disease control are defined as below:
  * Pre-DM: Reduction in HbA1c
  * HT: SBP/DBP < 140/90 millimetres of mercury (mmHg)
  * DM: HbA1c < 7%
The additional costs for delivering the CDCC Pilot Scheme by the costing questionnaire | 12 months
  The additional costs incurred on the CDCC Pilot Scheme from healthcare providers' perspective estimated from the manpower and pay scale of staff reported in the questionnaire, as well as the cost for acquiring physical space, equipment, and other IT infrastructure needed for the program. Costs will be presented as absolute values (HKD and USD).
The cost-effectiveness for delivering the CDCC Pilot Scheme on the incremental cost-effectiveness ratio | 12 months
  The incremental cost-effectiveness ratio (ICER) per individual achieving the target outcome of disease control for the CDCC Pilot Scheme compared to the cost-effectiveness threshold of 1 annual Gross Domestic Product (GDP) after 12 months

SECONDARY OUTCOMES:
Experience and satisfaction of CDCC participants by the experience and enablement questionnaire | Experience and satisfaction of CDCC participants will be evaluated at 3 months and 12 months after recruitment
  Participants' experience and satisfaction of services provided by the CDCC Pilot Scheme will be measured by self-reported experience and enablement questionnaire. It includes the standardized Patient Enablement Index with a total score ranging from 0 to 12, where higher scores indicate a better outcome. Other items were developed and adapted based on similar questionnaires. Patient experience and satisfaction levels will be assessed on a 4-point Likert scale with a higher score suggesting better satisfaction / experience.
Number of attendance to doctor consultation on times in comparison groups | 12 months
  Self-reported attendance to doctor consultation over the past 12 months for patients in comparison groups.
Rate of diagnosis of HT and/or DM on dichotomous yes/no response in comparison groups | 12 months
  Self-reported diagnosis of HT and/or DM on dichotomous yes/no response over the past 12 months for patients in comparison groups.
Changes in mean HbA1c/FPG in percent between two groups | 12 months
  Differences in the changes in mean HbA1c/fasting plasma glucose (FPG) from baseline to 12 months between pre-DM patients enrolled in the CDCC Pilot Scheme compared to comparison group.
Changes in mean SBP and DBP in millimeter of mercury between two groups | 12 months
  Differences in the changes in mean SBP and DBP from baseline to 12 months between hypertension patients enrolled in the CDCC Pilot Scheme and comparison group.
Changes in mean of HbA1c in percent between two groups | 12 months
  Differences in the changes in mean of HbA1c from baseline to 12 months between DM patients enrolled in the CDCC Pilot Scheme and comparison group.
Changes in BMI in kilogram per square metre between two groups | 12 months
  Differences in BMI from baseline to 12 months between patients enrolled in the CDCC Pilot Scheme compared to comparison group.
Changes in the rate of smoking cessation and rate of alcohol abstinence between two groups by the Health Risk Factor Assessment | 12 months
  Changes in the rate of smoking cessation and rate of alcohol abstinence between two groups by the Health Risk Factor Assessment
The predicted 10-year cardiovascular disease (CVD) risk between two groups | 12 months
  Differences in the predicted 10-year CVD risk using Framingham Risk Score and local CVD risk prediction model between patients enrolled in the CDCC Pilot Scheme compared to comparison group. The Framingham Risk Score ranges from 0% to 100% where higher scores indicate poorer outcomes.
Amount of direct medical costs between two groups | 12 months
  The direct medical costs of CDCC participants as compared with non-CDCC participants

CONTACTS AND LOCATIONS:
Locations (1):
- Jockey Club Building for Interdisciplinary Research 5 Sassoon Road, Pok Fu Lam, HONG KONG, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mak IL, Liu KSN, Wong ZCT, Xu VYH, Yu EYT, Ha TKH, Wong WCW, Tse ETY, Chan L, Ng APP, Choi EPH, Roland M, Bishai D, Lam CLK, Wan EYF. Evaluation of the effectiveness and cost-effectiveness of the chronic disease co-care (CDCC) Pilot Scheme: a study protocol. BMC Prim Care. 2025 Mar 19;26(1):73. doi: 10.1186/s12875-025-02765-6. PMID 40108515